CLINICAL TRIAL: NCT03634826
Title: A Prospective Study of Longitudinal Monitoring in Surgical Lung Cancer Patients by Circulating Tumor DNA and Its Methylation
Brief Title: Monitoring of Circulating Tumor DNA and Its Aberrant Methylation in the Surveillance of Surgical Lung Cancer Patients (MEDAL, MEthylation Based Dynamic Analysis for Lung Cancer).
Acronym: MEDAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1802
Record Dates: First submitted 2018-08-05; First posted 2018-08-17 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Carcinoma; Lung Cancer; NSCLC; Lung Neoplasm
Keywords: circulating tumor DNA; ctDNA methylation; lung cancer; surveillance
MeSH Terms: conditions — Carcinoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue and blood samples were collected from each patient. Time for blood sample collection: 1) Preoperation. 2) The 3rd day of postoperation. 3) Regular follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conduct a prospective study to confirm the value of circulating tumor DNA and its aberrant methylation in longitudinal monitoring of surgical lung cancer patients.

DETAILED DESCRIPTION:
Studies have already demonstrated the feasibility of circulating tumor DNA as a surrogate to reveal tumor mutation status in lung cancer patients and a few researches have shown the potential ability of using circulating tumor DNA in surveillance. However, no study focused on the value of methylation status of circulating tumor DNA in the surveillance and no strict prospective study has been performed in surgical lung cancer patients.

The investigators plan to analyze the dynamic change of circulating tumor DNA and its methylation status longitudinally from preoperation to long term follow-up in surgical lung cancer patients, and compare assessment value between circulating tumor DNA detection with methylation , traditional imaging examinations and traditional blood tumor markers in the monitoring process.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 80 years

* Lung cancer was suspected preoperatively.
* Received curative surgical therapy
* No malignant tumor history within the past 5 years
* No being received any treatment prior to resection
* Patients must have given written informed consent

Exclusion Criteria:

* The pulmonary nodule is pure ground glass opacity
* Unable to comply with the study procedure
* The postoperative pathology is not NSCLC.
* Unqualified blood samples

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed lung cancer patients who received surgical therapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between patients' recurrence and quantitative detection of circulating tumor DNA (ctDNA) concentration, including the quantitative detection of ctDNA mutations and ctDNA aberrant methylation. | 3 years

SECONDARY OUTCOMES:
The concordance of ctDNA genomic and methylation status alterations detected in peripheral blood samples with those in matched tumor samples. | 1 year
  Concordance will be defined as matched ctDNA and tumor DNA has the same identified mutations (methylation status alterations) or has no mutation (methylation status alteration). Concordance rate (%) will be calculated by consistent patient number and total patient number.
The variation of aberrant methylated ctDNA concentration before surgery, 3 days after surgery and 1 month after surgery. | 1 year
Correlation between disease free time and quantitative detection of ctDNA genomic alterations or methylation status alterations in patients who receives adjuvant therapy. | 3 years
Leading time of tumor relapse detection by circulating tumor DNA and methylation status than traditional radiological methods. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Study Chair — Peking University People's Hospital Thoracic Surgery Department
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen K, Kang G, Zhang Z, Lizaso A, Beck S, Lyskjaer I, Chervova O, Li B, Shen H, Wang C, Li B, Zhao H, Li X, Yang F, Kanu N, Wang J. Individualized dynamic methylation-based analysis of cell-free DNA in postoperative monitoring of lung cancer. BMC Med. 2023 Jul 14;21(1):255. doi: 10.1186/s12916-023-02954-z. PMID 37452374
- [Derived] Kang G, Chen K, Yang F, Chuai S, Zhao H, Zhang K, Li B, Zhang Z, Wang J. Monitoring of circulating tumor DNA and its aberrant methylation in the surveillance of surgical lung Cancer patients: protocol for a prospective observational study. BMC Cancer. 2019 Jun 13;19(1):579. doi: 10.1186/s12885-019-5751-9. PMID 31195991